CLINICAL TRIAL: NCT00409539
Title: A 10-week Randomised, DB, PG, PC Phase 2 Study to Investigate the Extent of Symptom Relief and the Safety and Tolerability of SMP-986 (20, 40, 80 and 120 mg) Administered Once Daily for 8 Weeks to Patients With Overactive Bladder Syndrome
Brief Title: SMP-986 Phase 2 Proof of Concept in Patients With Overactive Bladder Syndrome (OABS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Collaborators: Dainippon Sumitomo Pharma America (Industry); ICON Clinical Research (Industry); ClinPhone, Inc. (Industry); Covance (Industry); PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3601113
Record Dates: First submitted 2006-12-08; First posted 2006-12-11 (Estimated); Results first posted 2014-12-10 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Overactive Bladder Syndrome (OABS)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Placebo Comparator): Placebo run-in phase. 2 week duration.
  Interventions: Drug: Placebo
- 2 (Placebo Comparator): To be taken for the 8 week duration, in parallel with alternative arms (doses of 20, 40, 80 or 120mg SMP-986).
  Interventions: Drug: Placebo
- 3 (Experimental): 20mg dose of SMP-986 to be taken once daily for 8 week duration.
  Interventions: Drug: SMP-986
- 4 (Experimental): 40mg dose of SMP-986 to be taken for 8 week duration.
  Interventions: Drug: SMP-986
- 5 (Experimental): 80mg dose of SMP-986 to be taken for 8 week duration.
  Interventions: Drug: SMP-986
- 6 (Experimental): 120mg dose of SMP-986 to be taken for 8 week duration.
  Interventions: Drug: SMP-986

INTERVENTIONS:
Drug: Placebo — Placebo, 2 week duration.
  Arms: 1
Drug: Placebo — Taken for the 8 week duration, in parallel with alternative arms (doses of 20, 40, 80 or 120mg SMP-986).
  Arms: 2
Drug: SMP-986 — Comparison of varying dosages (20, 40, 80 or 120mg) of SMP-986 against placebo. Dosing is to occur once daily, in the morning, for a duration of 8 weeks
  Arms: 3; 4; 5; 6

SUMMARY:
SMP-986 is a compound being developed for the treatment of overactive bladder syndrome (OABS). This clinical study is designed to test the hypothesis that SMP-986 at doses of 20mg, 40mg, 80mg or 120mg provides greater symptom relief in OABS compared to placebo. The hypothesis will be tested by measuring the change in mean voids/24 hrs after treatment with SMP-986 compared to placebo, as well comparing the change in: the severity of urgency episodes, mean number of urgency episodes/24 hr, mean number of incontinence episodes/24 hr and the mean void volume/void between SMP-986 and placebo.

DETAILED DESCRIPTION:
A multicenter study conducted in patients with OABS comprising a 2-week single blind placebo run-in period followed by an 8-week randomized, double-blind, placebo controlled treatment period with patients randomized to receive 20 mg, 40 mg, 80 mg or 120 mg SMP 986 or placebo in a 1:1:1:1:1 ratio in parallel groups on an outpatient basis with study center visits.

ELIGIBILITY:
Inclusion Criteria:

Main Inclusion Criteria:

* Males, or females who are not of child-bearing potential
* Aged 20-80 years (inclusive) with a diagnosis of OABS based on symptomatic reporting over a period of 6 months (micturition frequency, and urgency with or without incontinence) prior to screening.

Exclusion Criteria:

Main Exclusion Criteria:

* Patients will be excluded if there is an indication of any bladder outlet obstruction or polyuria
* Patients with the following conditions, or who have undergone the following procedures, will be excluded:

  * stress urinary incontinence
  * pelvic organ prolapse ( stage 2)
  * genitourinary or lower bowel surgery (within 12 months prior to screening),
  * pathological conditions including poorly controlled diabetes, painful bladder syndrome/interstitial cystitis or history of chronic urinary tract infection
  * neurological conditions including multiple sclerosis, Parkinson's disease or neuropathy)
* Patients will also be excluded if they have an indwelling catheter or perform intermittent self catheterisation
* Patients should not have a current or past medical condition contraindicating the use of antimuscarinics and must have discontinued use of the following drugs:

  * drugs used to treat OABS or urinary incontinence
  * cholinergics
  * anticholinergics
  * alpha adrenergic antagonists
  * opioid analgesics
  * compound analgesics containing an opioid
  * warfarin
* Patients with a current or past malignancy (within the last 5 years)
* Patients who have ever had a tumour affecting the genitourinary tract (not including benign prostatic hyperplasia) will be excluded.
* Patients will be ineligible if they have a clinically significant cardiac, neurological, hepatic, renal, respiratory, haematological or gastrointestinal disorder (including, a significant history of constipation or an active bowel disease e.g. inflammatory bowel disease) or any other illness which in the opinion of the Investigator would preclude the safe or compliant participation of a subject.
* Patients will be excluded if they are unable to complete the study diary

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2006-12; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof C Chappel, Principal Investigator — Royal Hallamshire Hospital
Locations (68):
- United States (21):
  - Visions Clinical Research, Tuscon, Arizona
  - Peninsula Urology Center, Atherton, California
  - San Bernadino Urological Association Medical Group, San Bernadino, California
  - 9040 Friars Road, San Diego, California
  - South Florida Medical Research, Aventura, Florida
  - Visions Clinical Research, Boynton Beach, Florida
  - Florida Healthcare Research, Ocala, Florida
  - Southern Research Group, Centre Point Boulevard, Tallahassee, Florida
  - Atlanta Medical Research, Alpharetta, Georgia
  - Urological Surgeons of IL, Kankakee, Illinois
  - Regional Urology, Shreveport, Louisiana
  - Accumed Research Associate, Garden City, New York
  - Hudson Valley Urology, Kingston, New York
  - New York Urological Associates, PC, New York, New York
  - Hudson Valley Urology, Poughkeepsie, New York
  - Unifour Medical Research, Hickory, North Carolina
  - University of Pittsburg, Dept Urology, Pittsburgh, Pennsylvania
  - Volunteer Research Group, Knoxville, Tennessee
  - 5920 Saratoga Boulevard, Corpus Christi, Texas
  - National Clinical Research Inc, Richmond, Virginia
  - 801 W. 5th Avenue, Spokane, Washington
- Estonia (3):
  - East Tallinn Central Hospital, Tallinn
  - West Tallinn Central Hospital, Tallinn
  - Tartu University Clinic, Tartu
- France (3):
  - Hopital Rothschild, Paris
  - Hopital Tenon, Paris
  - Hopital Rangueil - CHU Toulouse, Toulouse
- Germany (15):
  - Gem. Praxis fur Urologie und Mannerheilkunde, Berlin
  - Klinische Forschung Berlin, Berlin
  - Urologische Praxis, Berlin
  - Urologische Praxis, Buchholz
  - Gem. Praxis Jacobi & Hellmis, Duisburg
  - Urologische Gem. Praxis, Düsseldorf
  - Urologische Praxis, Düsseldorf
  - Poststr. 25, Hagenow
  - Urologische Gem. Praxis, Hamburg
  - Urologische Praxisgemeinschaft, Hamburg
  - Urologische Praxis, Leipzig
  - Universitat Heidelberg, Mannheim
  - HauptstraBe 10, Markkleeberg
  - Josef-Retzer-Str. 46, München
  - Beckenboden Zentrum Munchen, München
- Latvia (2):
  - Medical Company ARS, Riga
  - P. Stradins Hospital, Riga
- Lithuania (3):
  - Kaunas 2nd Clinical Hospital, Kaunas
  - Kaunas Hospital, Kaunas
  - Vilnius Santariskes Clinics, Vilnius
- Poland (11):
  - Oddzial Urologii, Bydgoszcz
  - Akdemickie Centrum Kliniczne, Gdansk
  - Medical University of Selesia, Katowice
  - Non-public Healthcare Unit, Kutno
  - UI.G. Narutowicza 28, Lodz
  - Instytut Zdrowia Matki Polki, Lodz
  - University School of Medicine, Lublin
  - Clinical Dept of Urology, Medical Postgraduate Education, Warsaw
  - Military Institute of Medicine, Warsaw
  - Klinika Urologii Akademii, Warsaw
  - Ackademicki Szpital Klniczny, Wroclaw
- Spain (5):
  - Hospital Universitario, Santa Cruz de Tenerife, Canary Islands
  - Hospital De Terrassa, Barcelona
  - Servicio de Ginecologia, Barcelona
  - Hospital Sant Joan De Deu, Barcelona
  - Fundacion Hospital Alcorcon, Madrid
- United Kingdom (5):
  - Aberdeen Royal Infirmary, Aberdeen
  - Addenbrooke's Hospital, Cambridge
  - Leighton Hospital, Crewe
  - King's College Hospital, London
  - The Royal Hallamshire Hospital, Sheffield

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 550 subjects were enrolled into the 2 week placebo run-in phase prior to randomization.
Groups:
- Placebo: Placebo run-in phase. 2 week duration.
  Placebo: Placebo, 2 week duration.
- 20mg Dose of SMP-986: 20mg dose of SMP-986 to be taken once daily for 8 week duration.
  SMP-986: Comparison of varying dosages (20, 40, 80 or 120mg) of SMP-986 against placebo. Dosing is to occur once daily, in the morning, for a duration of 8 weeks
- 40mg Dose of SMP-986: 40mg dose of SMP-986 to be taken for 8 week duration.
  SMP-986: Comparison of varying dosages (20, 40, 80 or 120mg) of SMP-986 against placebo. Dosing is to occur once daily, in the morning, for a duration of 8 weeks
- 80mg Dose of SMP-986: 80mg dose of SMP-986 to be taken for 8 week duration.
  SMP-986: Comparison of varying dosages (20, 40, 80 or 120mg) of SMP-986 against placebo. Dosing is to occur once daily, in the morning, for a duration of 8 weeks
- 120mg Dose of SMP-986: 120mg dose of SMP-986 to be taken for 8 week duration.
  SMP-986: Comparison of varying dosages (20, 40, 80 or 120mg) of SMP-986 against placebo. Dosing is to occur once daily, in the morning, for a duration of 8 weeks
Period: Overall Study
Arm/Group | Placebo | 20mg Dose of SMP-986 | 40mg Dose of SMP-986 | 80mg Dose of SMP-986 | 120mg Dose of SMP-986
Started | 111 | 111 | 109 | 109 | 110
Completed | 100 | 100 | 95 | 97 | 85
Not Completed | 11 | 11 | 14 | 12 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 20mg Dose of SMP-986 | 40mg Dose of SMP-986 | 80mg Dose of SMP-986 | 120mg Dose of SMP-986 | Total
Number analyzed (Participants) | 111 | 111 | 109 | 109 | 110 | 550
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (11.15) | 62.0 (9.60) | 61.5 (9.93) | 61.6 (9.04) | 61.1 (10.08) | 61.4 (9.96)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 64 | 63 | 66 | 63 | 65 | 321
  >=65 years | 47 | 48 | 43 | 46 | 45 | 229
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 92 | 89 | 93 | 95 | 465
  Male | 15 | 19 | 20 | 16 | 15 | 85
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 1 | 1 | 6 | 14
  White | 107 | 108 | 107 | 106 | 103 | 531
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 23 | 14 | 15 | 25 | 103
  Poland | 31 | 27 | 32 | 30 | 30 | 150
  Germany | 29 | 35 | 40 | 39 | 30 | 173
  Estonia | 4 | 5 | 2 | 6 | 6 | 23
  France | 1 | 1 | 0 | 1 | 1 | 4
  Latvia | 7 | 8 | 6 | 7 | 10 | 38
  Lithuania | 11 | 5 | 13 | 7 | 3 | 39
  Spain | 2 | 3 | 1 | 1 | 5 | 12
  United Kingdom | 0 | 4 | 1 | 3 | 0 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 8 in the Number of Voids/24 Hours
Time Frame: 8 Weeks
Measure: Least Squares Mean (Standard Error); unit: voids/24 hrs.
Arm/Group | Placebo | 20mg Dose of SMP-986 | 40mg Dose of SMP-986 | 80mg Dose of SMP-986 | 120mg Dose of SMP-986
Number analyzed (Participants) | 111 | 111 | 109 | 109 | 110
voids/24 hrs. | -1.06 (2.223) | -1.44 (2.402) | -1.78 (2.376) | -2.41 (2.383) | -1.92 (2.145)

2. Secondary Outcome: To Assess the Safety and Tolerability of 20, 40, 80 and 120 mg SMP 986 (o.d) Following 8-weeks of Treatment in Patients With Over Active Bladder Syndrome
Description: Treatment emergent adverse event summary
Time Frame: 8 Weeks
Measure: Number; unit: participants
Arm/Group | Placebo | 20mg Dose of SMP-986 | 40mg Dose of SMP-986 | 80mg Dose of SMP-986 | 120mg Dose of SMP-986
Number analyzed (Participants) | 111 | 111 | 109 | 109 | 110
participants | 61 | 62 | 61 | 87 | 90

ADVERSE EVENTS:
Time Frame: 8 Weeks
Arm/Group | Placebo | 20mg Dose of SMP-986 | 40mg Dose of SMP-986 | 80mg Dose of SMP-986 | 120mg Dose of SMP-986
Serious Adverse Events (participants affected / at risk) | 0/111 | 1/111 | 1/109 | 0/109 | 3/110
Other Adverse Events (participants affected / at risk) | 39/111 | 40/111 | 50/109 | 78/109 | 81/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=111) | 20mg Dose of SMP-986 (N=111) | 40mg Dose of SMP-986 (N=109) | 80mg Dose of SMP-986 (N=109) | 120mg Dose of SMP-986 (N=110)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Loss of Conciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=111) | 20mg Dose of SMP-986 (N=111) | 40mg Dose of SMP-986 (N=109) | 80mg Dose of SMP-986 (N=109) | 120mg Dose of SMP-986 (N=110)
Vision Blurred (Eye disorders) | 0 (0) | 1 (1) | 2 (2) | 7 (7) | 5 (5)
Abdominal Pain Upper (Gastrointestinal disorders) | 2 (2) | 6 (6) | 2 (2) | 3 (3) | 3 (5)
Constipation (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1) | 8 (8) | 10 (10)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 4 (4) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 13 (13) | 22 (25) | 35 (39) | 64 (70) | 74 (80)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 5 (6) | 6 (6) | 3 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 4 (4)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 4 (4) | 2 (2)
Nasopharyngitis (Infections and infestations) | 7 (7) | 4 (4) | 4 (4) | 4 (4) | 4 (4)
Urinary Tract Infection (Infections and infestations) | 6 (6) | 3 (3) | 3 (3) | 6 (6) | 3 (6)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 5 (22) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 9 (12) | 6 (9) | 5 (7) | 10 (12) | 7 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In addition to the <60-180 day restriction above, since this is a multicenter study, 1st publication of study results shall be made with other participating study sites as a multicenter publication; provided, if a multicenter publication is not forthcoming within 24 months following completion of study at all sites, the PI shall be free to publish.